CLINICAL TRIAL: NCT07386418
Title: Study of Lesion-Specific Invasive Haemodynamic Angina Thresholds
Acronym: ORBITA-SOLAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); University Hospitals Dorset NHS Foundation Trust (Other Government); Mid and South Essex NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 199514
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Angina (Stable); Ischaemic Heart Desease; Coronary Artery Disease(CAD)
Keywords: Angina; Coronary physiology; Coronary haemodynamics; Placebo-control; Symptoms
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Angina Pectoris | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: All participants will partake in the same research protocol.
Masking Description: During cardiac catheterisation, there will be one blinded component to verify the reproducibility of symptoms against placebo. One true and one placebo balloon inflation will be performed, in a randomised order. Both the participant and outcome assessor will be blinded to the order of true or placebo balloon inflation. The participant will be asked to report any symptoms they have.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with stable coronary artery disease (Experimental): 1. Symptoms of stable angina
  2. Evidence of ischaemia on an invasive or non-invasive test
  3. Two coronary stenoses amenable to percutaneous coronary intervention (PCI)
  Interventions: Procedure: Percutaneous coronary intervention (PCI); Diagnostic Test: Measurement of the angina threshold

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Clinically indicated PCI for the management of stable angina
Diagnostic Test: Measurement of the angina threshold — Following stenting, the order in which to perform the angina threshold assessment at the location of each stent will be randomised. A non-compliant balloon with gradually be inflated over a pressure wire within the deployed stent to re-introduce stenosis. Simultaneously, the participant will exercise on a supine ergometer. At the point when angina is reproduced, the patient will rest and further balloon inflation will stop. Physiological measurements using the pressure wire will be taken with the inflated balloon in situ. This will represent the invasive physiological angina threshold. The balloon will then be deflated and removed. These steps will be repeated at the location of the second stent.

SUMMARY:
ORBITA-SOLAR is an invasive physiological cardiac catheterisation study that aims to determine whether different coronary stenoses have different angina thresholds. The angina threshold is defined as the amount of coronary flow reduction required to reproduce symptoms. Sixty patients with symptoms of stable angina and 2 coronary artery stenoses amenable to percutaneous coronary intervention (PCI) will be recruited. This study will use intra-coronary balloon inflation during supine exercise on an ergometer to measure the fractional flow reserve (FFR) and non-hyperemic pressure ratio (NHPR) that relates to angina onset, in real time, at the location of each stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility for PCI due to angina or angina-equivalent symptoms on exertion
2. 2 severe epicardial stenoses in a major coronary artery, defined as:

   1. ≥70% stenosis in a coronary artery with ≥2.5mm diameter, on invasive coronary angiography (ICA)
   2. Severe stenosis in a vessel with ≥2.5mm diameter, on CTCA
3. Evidence of ischaemia on an invasive or non-invasive test, including:

   1. Physiological test during invasive coronary angiography (ICA)
   2. Dobutamine stress echocardiography (DSE)
   3. Stress perfusion cardiac magnetic resonance (CMR)
   4. Myocardial perfusion scintigraphy (MPS)
   5. Fractional flow reserve computed-tomography (FFR-CT)

Exclusion Criteria:

1. Age <18 years
2. Acute coronary syndrome within 3 months
3. Previous coronary artery bypass graft
4. Significant left main stem disease
5. Single lesion amenable to PCI
6. Chronic total occlusion of the target artery
7. Moderate to severe valve disease
8. LVEF ≤40%, contraindication to PCI or drug-eluting stents
9. PCI performed with drug-eluting balloons without stenting
10. Contraindication to antiplatelet therapy
11. Contraindication to adenosine
12. Physical inability to exercise with an ergometer
13. Femoral artery access
14. Pregnancy
15. Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Intra-individual difference in FFR and NHPR angina thresholds | Intra-procedural
  Difference in invasively measured physiological angina thresholds at the site of the 2 stents within each participant, stratified by vascular territory and lesion location along a vessel.

SECONDARY OUTCOMES:
Correlation of the angina threshold with other invasive physiological assessments | Intra-procedural
  Including coronary artery disease pattern (focal, diffuse or mixed), presence of microvascular disease (IMR and CFR), extent of collateral flow (CFI), and pre- and post-PCI ischaemia (FFR and RFR)
Correlation of the angina threshold with anatomical characteristics assessed with computed tomography coronary angiography (CTCA) | 14 days
  Including proportion of myocardial mass subtended (%), coronary artery territory (LAD, LCx, RCA), and lesion location along a vessel (proximal, mid, distal)
Correlation of the angina threshold with anatomical characteristics assessed with quantitative coronary angiography (QCA) | 14 days
  Including lesion length (mm), minimum lumen diameter, (mm) percent diameter stenosis (%), and reference vessel diameter (mm)
Correlation of the angina threshold with anatomical characteristics assessed with intravascular imaging | Intra-procedural
  Including lesion length (mm), pre-PCI minimum lumen area (mm2), post-PCI minimum stent area (mm2), reference vessel cross-sectional area (mm2), plaque characteristics (lipid, fibrotic, calcific)
Correlation of the angina threshold with features on a stress perfusion cardiac magnetic resonance imaging (CMR) scan | 14 days
  Including myocardial perfusion reserve (MPR), number of segments of infarcted myocardium, and percentage mural infarct depth (%)
Correlation of the angina threshold with baseline symptoms, quality of life and pain perception | 14 days
  Assessed with the ORBITA-app and validated questionnaires (SAQ, EQ5D5L)

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Mid and South Essex NHS Foundation Trust, Basildon
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth
  - Imperial College Healthcare NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Portsmouth Hospitals University NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No